CLINICAL TRIAL: NCT05233514
Title: Effect of Aerobic Exercise on Inflammatory Markers in Polycystic Ovary Syndrome
Brief Title: Effect of Aerobic Exercise on Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, Professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POV
Record Dates: First submitted 2022-01-29; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: participants were divided into two groups equal in number: the aerobic exercise group (AEM), and the Metformin group (M). The AEM group performed aerobic exercise three times a week for 12 weeks in addition to Metformin treatment. The M group received Metformin only
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (AEM) (Experimental): The AEM group performed aerobic exercise three times a week for 12 weeks in addition to Metformin treatment.
  Interventions: Other: Aerobic exercise in addition to Metformin treatment
- Metformin group (M) (Active Comparator): The M group received Metformin only
  Interventions: Other: Aerobic exercise in addition to Metformin treatment

INTERVENTIONS:
Other: Aerobic exercise in addition to Metformin treatment — The aerobic exercises were walking on the treadmill for 30 minutes at a 0% slope, including three phases: the warming-up phase, which consisted of walking on the treadmill for five minutes at low intensity (30% of Maximum Heart Rate, MHR), the actual phase, which consisted of walking on the treadmill for 20 min at moderate intensity (60 -70% of MHR) and the cooling phase, which consisted of walking on the treadmill for five minutes at low intensity (30% of MHR). The MHR was calculated according to the equation (210- age in years). Both the AEM and M groups received metformin 1,500 mg daily for a further 12 weeks.

SUMMARY:
The development of Polycystic Ovary Syndrome has been linked to chronic low-grade inflammation (PCOS). In this context, the current study looked into the effects of aerobic exercise on IL6, TNF, and C-reactive protein (CRP) in PCOS women. This was a randomized clinical trial including 40 females diagnosed with PCOS who were between the ages of 25 and 35. The participants were divided into two groups, each with an equal number of individuals: aerobic exercise (AEM) and Metformin (M). At baseline and after 12 weeks of intervention, participants' levels of IL6, TNF, and CRP were measured.

ELIGIBILITY:
Inclusion Criteria:

* Mean age of 26.7 ± 2.3, body mass index (BMI) 23.6±3.5 kg/m2) .
* confirmation by medical history of hyperandrogenic oligo amenorrhea (<8 menses per year)
* PCO on ultrasonography of more than 10 ovarian follicles 2-9 mm in diameter

Exclusion Criteria:

* Disorders known to cause hyperandrogenisms, such as congenital adrenal hyperplasia, thyroid dysfunction, and hyperprolactinemia.
* Renal or hepatic dysfunction

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Level of Interleukin 6 | 12 weeks
Level of TNF-α | 12 weeks
level of C- reactive protein | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No